CLINICAL TRIAL: NCT04461158
Title: Utilizing a Lupus Patient Navigator Program (LPNP) to Address Barriers to Care Related to Access to Preventive and Specialty Healthcare, Medication Adherence and Health Literacy in Systemic Lupus Erythematosus (SLE) for Minority Patients
Brief Title: CCCR Lupus Patient Navigator Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); University of Alabama at Birmingham (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 00095036; 3P30AR072582-03S1 (NIH)
Record Dates: First submitted 2020-07-01; First posted 2020-07-08 (Actual); Results first posted 2024-08-06 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Systemic Lupus Erythematosus (SLE)
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional Group (Experimental)
  Interventions: Behavioral: Patient Navigator Services

INTERVENTIONS:
Behavioral: Patient Navigator Services — The navigator services most commonly provided include facilitation and coordination of care, practical support, including transportation and financial assistance, appointment scheduling and reminders, education and psychosocial support

SUMMARY:
To address the health disparities in SLE outcomes for minorities, targeted intervention will be used to address the common barriers to care among patients; a comprehensive patient navigator approach will be utilized based on evidence from prior studies is the purpose of this research. The navigator services most commonly provided include facilitation and coordination of care, practical support, including scheduling transportation and referrals to financial assistance programs, appointment scheduling and reminders, education and psycho-social support. The most effective patient navigators address both health system and patient barriers.

ELIGIBILITY:
Inclusion Criteria:

1. Self-identified Minority.
2. Patients ≥ 18 years of age as documented in the electronic medical record.
3. Meeting either American College of Rheumatology or SLICC Classification Criteria for SLE as documented in the electronic medical record.
4. Ability to speak and understand English by self-report.
5. In the past six months having ≥ 1 missed clinic or diagnostic study/laboratory visit as documented in the electronic medical record, or self-reported failure to adhere with prescribed medical therapy for SLE.
6. In the past six months having been prescribed at least one immunosuppressive medication for SLE activity as documented in the electronic medical record regardless of whether taking the medication.
7. Currently enrolled into the Core Center for Clinical Research (CCCR; Pro 00021985) with properly executed Informed Consent Document and HIPAA Authorization.
8. Have telephone access.

Exclusion Criteria:

1. Unwilling or unable to give informed consent.
2. Being a prisoner or institutionalized individual.
3. Without telephone access.
4. Do not meet all of the inclusion criteria listed above.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2020-09-03 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jim C. Oates, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Usual Care Comparison Group: Usual Care Comparison Group meeting eligibility criteria for intervention but not receiving Lupus Patient Navigator Program services.
Period: Overall Study
Arm/Group | Interventional Group | Usual Care Comparison Group
Started | 52 | 23
Completed | 46 | 23
Not Completed | 6 | 0

BASELINE CHARACTERISTICS:
Population: Patients with SLE
Groups:
- Intervention Group: Receiving Lupus Patient Navigator Program services.
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Usual Care Comparison Group | Total
Number analyzed (Participants) | 52 | 23 | 75
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 52 | 23 | 75
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.0 (11.4) | 34.8 (10.6) | 34.2 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 18 | 68
  Male | 2 | 5 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 49 | 21 | 70
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 50 | 22 | 72
  White | 2 | 0 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 52 | 23 | 75
Age at lupus onset [Mean (Standard Deviation); unit: years] | 25.6 (10.2) | 28.4 (10.3) | 26.5 (10.2)

OUTCOME MEASURES:

1. Primary Outcome: Improvement in Quality of Life
Description: Qualify of life measured by the "LupusPRO" patient-reported questionnaire administered at Baseline and 12 Months in the Intervention Group, resulting in a LupusPRO score.
  LupusPRO (v1.8) includes 43 items with domains of Lupus Symptoms, Lupus Medication, Physical Health, Emotional Health, Pain, Sleep, Procreation, Cognition, Body Image, Desires-Goals, Coping, Social Support and Satisfaction with Care rated on a 5 point Likert scale, where 0=None of the time/not applicable, 1= A little of the time, 2= Some of the time, 3=Most of the time, 4= All of the time, 5= Not applicable.
  Total scores measure health (HRQOL) and non-health related quality of life (Non HRQOL). Item scores are totaled for each domain item and the mean domain score is obtained by dividing the total score by the number of items in that domain. The mean raw domain score is transformed to scores ranging from 0 (worst QOL) to 100 (best QOL) by dividing by 4 (the number of Likert responses {5 responses
Time Frame: 12 months - from baseline to 12 month visit
Population: 52 patients with SLE self identified as a minority, met inclusion / exclusion criteria, and provided informed consent to participate with the Lupus Patient Navigator Program intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Interventional Group
Number analyzed (Participants) | 52
score on a scale
  Baseline Health-related QOL | 59.2 (20.6)
  12 Month Health-related QOL: number analyzed (Participants) | 46
  12 Month Health-related QOL | 63.6 (22.1)

2. Secondary Outcome: Improvement in Medication Adherence
Description: Adherence with prescribed medical therapies will be defined as the ratio between the number of therapy-days supplied to the number of days until the prescription was refilled and compared between Lupus Patient Navigator Program (LPNP) participants and usual care patients. Medication adherence rates will be estimated by charts review and comparing these medications to pharmacy records on dates and quantities filled. Included medication classifications will include antihypertensives, immunosuppressants, Plaquenil (hydroxychloroquine), and glucocorticoids. Additionally, overall pill burden will be compared between LPNP participants and usual care patients. LPNP participants' medication diaries will be reviewed to determine self-reported adherence.
Time Frame: 12 months - from baseline to 12 month visit
Reporting Status: Not Posted, anticipated posting 2025-08

3. Secondary Outcome: Improvement in Patient-reported Lupus-specific Disease Status
Description: Changes in patient-reported lupus-specific disease status (measured by the LupusPRO v1.7) over time, from Baseline, 3, 6, 9, and 12 months, compared between interventional and usual care groups will be completed at the start and end of participation. The LupusPRO is a validated, comprehensive patient reported quality of life questionnaire specific for patients with lupus. Domain areas include: lupus symptoms, cognition, physical health, pain vitality, procreation, emotional health, body image, desires-goals, social support, coping, and satisfaction with care.
Time Frame: 12 months - from baseline to 12 month visit
Reporting Status: Not Posted, anticipated posting 2025-08

4. Secondary Outcome: Improvement in Adherence With Medical Providers and Services
Description: Adherence with medical providers and services will be the ratio of number of visits scheduled to the number of visits kept. Rates will be compared between LPNP participants and usual care patients.
Time Frame: 12 months - from baseline to 12 month visit
Reporting Status: Not Posted, anticipated posting 2025-08

ADVERSE EVENTS:
Time Frame: 1 year
Description: Only deaths were assessed. Serious and non-serious/other adverse events were not assessed. Patients are already routinely monitored by their clinicians for standard of care.
Arm/Group | Interventional Group | Usual Care Comparison Group
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-02-04): https://cdn.clinicaltrials.gov/large-docs/58/NCT04461158/Prot_SAP_001.pdf
  • Informed Consent Form (2020-10-07): https://cdn.clinicaltrials.gov/large-docs/58/NCT04461158/ICF_000.pdf